CLINICAL TRIAL: NCT00654212
Title: Endo-Laparoscopic Approach Versus Conventional Open Surgery in the Management of Obstructing Left-sided Colon Cancer: A Randomized Trial
Brief Title: Endo-Laparoscopic Approach Versus Conventional Open Surgery in Obstructing Left-sided Colon Cancer: RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Cheung Yui Shan, Consultant Surgeon, Pamela Youde Nethersole Eastern Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shan
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Colonic Neoplasms
Keywords: stenting, laparoscopic surgery, colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Laparotomy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): endoluminal stenting followed by laparoscopic resection (endo-laparoscopic limb, the study group)
  Interventions: Procedure: endo-laparoscopic approach
- 2 (Other): emergency open surgery (open limb, the control group)
  Interventions: Procedure: open approach

INTERVENTIONS:
Procedure: endo-laparoscopic approach — endoluminal stenting followed by laparoscopic resection
  Other Names: Wallstent Enteral Endoprosthesis
  Arms: 1
Procedure: open approach — emergency open surgery
  Other Names: laparotomy
  Arms: 2

SUMMARY:
Objective: Whether temporary endoscopic decompression by Self-expanding metal stents (SEMS) could allow these patients to undergo successful laparoscopic resection (endo-laparoscopic approach) has never been previously studied. This randomized trial aims to compare this approach with emergency open surgery in the management of obstructing left-sided colon cancer.

DETAILED DESCRIPTION:
Introduction:

First reported in 1991, laparoscopic assisted colectomy is increasingly practised world-wide. Abundant evidence exists in the literature suggesting laparoscopic assisted colectomy, when compared with its open counterpart, is associated with more favourable short-term outcomes, better cosmesis, and better patient's satisfaction. Moreover, recent reports from large-scale randomized trials support the use of this minimally invasive technique in the treatment of colorectal cancer, a malignant condition common in many parts of the world. However, around 8-29% of patients with colorectal cancer present as acute large bowel obstruction, a condition used to be considered as a contraindication to laparoscopic surgery due to poor exposure and potential hazard of injury to the distended bowel. Thus, most cases of malignant large bowel obstruction mandate an emergency open surgery to relieve the obstruction and resect the tumour, with many patients, especially those with obstructing left-sided colon cancer, ending up with temporary or permanent stoma which can adversely affect their health-related quality of life.

Self-expanding metal stents (SEMS) was first described by Dohmoto in 1991 as an endoscopic palliative alternative for treating inoperable colon cancer. Three years later, Tejero et al. published a preliminary report of using SEMS as a 'bridge' to surgery in two patients with colonic obstruction 13. Since then, a number of publications as well as systemic review have shown that endoluminal stenting is a relatively simple and safe alternative to standard surgical management of acute malignant obstruction of the left colon, thereby obviating the need of emergency surgery or colostomy. However, whether temporary endoscopic bowel decompression by SEMS could allow patients with malignant left colonic obstruction to undergo successful laparoscopic resection (endo-laparoscopic approach) has never been studied in detail before. We therefore conducted the current trial to study the outcomes of this endo-laparoscopic approach in patients with obstructing left-sided colon cancer.

Patients and Methods:

This study is a randomized controlled trial designed to evaluate the outcomes of the endo-laparoscopic approach for patients with obstructing left-sided colon cancer, using patients undergoing emergency open surgery as controls. Only patients with obstructing left-sided colon cancer were studied because of the reported high incidence of stoma creation in this condition10,11, and because a homogeneous group of patients could be ensured to facilitate comparison of the two different approaches. A single surgical team consisting of two surgeons (C.C.C. and M.K.W.L.) and one camera assistant in the case of laparoscopic resection performed all operations with the patient under general anesthesia. The study was approved by the hospital ethical committee and was not supported by any commercial funds or sponsorship.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients (aged 18 or above) presenting with clinical features of left colonic obstruction were potential candidates.
* In the absence of peritonitis, right lower quadrant tenderness or grossly distended caecum (10cm or above in maximal dimension) on plain abdominal radiograph, an urgent water-soluble single contrast enema was performed to determine the level of obstruction within 24 hours of admission.
* Patients were recruited if the lower border of an obstructing tumour was found between the splenic flexure and rectosigmoid junction.
* Informed consent was obtained from every patient recruited in the trial.

Exclusion Criteria:

* Patients who did not give informed consent
* Patients who were considered unfit for operative treatment
* Patients with previous laparotomy
* Patients with clinically palpable tumor on abdominal examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-01; Primary Completion 2005-05 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
successful one-stage operation | till end of the study

SECONDARY OUTCOMES:
cumulative operative time, cumulative blood loss, conversion rate, post-operative pain, cumulative length of hospital stay, operative mortality, post-operative complications, ates of permanent stoma creation,disease recurrence, survival | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Li Ka Wah, FRCSEd, Study Director — PamelaNEH
Locations (1):
- Pamela Youde Nethersole Eastern Hosptial, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Cheung HY, Chung CC, Tsang WW, Wong JC, Yau KK, Li MK. Endolaparoscopic approach vs conventional open surgery in the treatment of obstructing left-sided colon cancer: a randomized controlled trial. Arch Surg. 2009 Dec;144(12):1127-32. doi: 10.1001/archsurg.2009.216. PMID 20026830